CLINICAL TRIAL: NCT01282788
Title: A Novel Sustainable Complementary Feeding Product for Infants and Young Children in the Democratic Republic of Congo: Caterpillar Cereal
Brief Title: Efficacy of Caterpillar Cereal for Complementary Feeding in the Democratic Republic of Congo
Acronym: CAT02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kinshasa School of Public Health (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Carl Bose, MD, Prinicipal investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-2071
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Malnutrition; Stunting of Growth; Iron Deficiency Anemia; Neurodevelopmental Impairment; Infectious Diseases Morbidity
Keywords: infant nutrition; complementary feeding; malnutrition; stunting of growth
MeSH Terms: conditions — Malnutrition; Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Diet (No Intervention): Infants in communities randomized to the traditional diet arm will not receive food supplements.
- Cereal (Experimental): All infants in communities randomized to the Cereal Arm will receive caterpillar cereal from 6-18 months of age.
  Interventions: Dietary Supplement: Caterpillar Cereal

INTERVENTIONS:
Dietary Supplement: Caterpillar Cereal — Infants will receive once-daily servings of caterpillar cereal (30 g from 6-12 months of ages and 45 g from 12-18 months of ages). Study food will be delivered to homes weekly by Community Coordinators, who will also observe feedings of the cereal during the home visit. Feedings will be observed 3x/week for the first 3 weeks after enrollment, then 1x/week until 18 months of age. Parents and other care providers will receive specific instructions about cereal preparation and general education about feeding practices, food preparation and hygiene. This information will be reinforced during weekly visits.
  Arms: Cereal

SUMMARY:
Two in every three infants in rural areas of the Democratic Republic of Congo (DRC) suffer from stunting of linear growth by 12 months of age. Stunting presumably results from breast milk supplementation after 6 months of age with complementary foods (CF) that provide inadequate protein and micro-nutrients. Although supplementation with selected micro-nutrients may avoid certain deficiency states, CF with animal source foods may be necessary to avoid stunting. Meat is not readily available in many Central African countries. However caterpillars, which are locally available and abundant, are a common staple in adult diets and may be a suitable substitute for animal source proteins in CF. The investigators developed a cereal made from dried caterpillars that has a nutrient content that appears to be ideal for CF and demonstrated maternal and infant acceptability. This study will investigate the efficacy in prevention of stunting of growth resulting from inadequate complementary foods.

A sub-study will evaluate the biologic effects of the caterpillar cereal to determine whether caterpillar cereal prevents iron deficiency anemia, reduces the incidence of neurodevelopmental impairment or infectious diseases.

DETAILED DESCRIPTION:
A randomized, controlled trial will be conducted in the Equateur Province. The study will be a cluster randomized, non-masked controlled trial of a daily intake of caterpillar cereal (Cereal Arm) versus the usual diet provided by the family (Traditional Diet Arm) from 6 to18 months of age. Eight communities (clusters) will be randomized to either the Cereal Arm or the Traditional Diet Arm of the study. A community will be comprised of approximately 10 to 12 rural villages served by one Health Center. Each Cereal community will be paired with a Traditional Diet community.

Educational Information

All participants will be provided with general education that will include: 1) critical messages about infant feeding and 2) instruction about hand hygiene and food preparation. The primary educators will be the Community Coordinators (CCs; specially-trained research nurses) working with the Health Center nurses. Messages will be delivered and reinforced with pictorial aids. Mothers in both arms will receive three repetitive messages to reinforce selected features of World Health Organization (WHO) recommendations for complementary feeding:

1. Feed thickened gruel or cereals every day
2. Feed infant/toddler at least 3 times a day
3. Maximize local food diversity

Cereal Arm All infants in communities randomized to the Cereal Arm will receive once-daily servings of caterpillar cereal (30 g from 6-12 months of ages and 45 g from 12-18 months of ages). Study food will be delivered to homes weekly by CCs, who will also observe feedings of the cereal during the home visit. Feedings will be observed 3x/week for the first 3 weeks after enrollment, then 1x/week until 18 months of age. Parents and other care providers will receive specific instructions about cereal preparation and general education about feeding practices, food preparation and hygiene. This information will be reinforced during weekly visits.

Traditional Diet Arm Infants in communities randomized to the Traditional Diet Arm will not receive food supplements. Parents and other care providers in this arm of the study will receive general education about feeding practices, food preparation and hygiene, with weekly reinforcement.

Study Population A total of 220 infants (approximately 27 from each community; 110 infants in each arm) will be enrolled in the study. Records of all births within study communities will be obtained from local Health Center records. When infants reach 5 months of age, caregivers of randomly selected infants will be approached by CCs to seek consent for participation in this study. They will be supported by the Provincial Coordinator (the physician who oversees community-based studies conducted by the Kinshasa School of Public Health-University of North Carolina Partnership) who will hold group information meetings to introduce the study to community leaders.

ELIGIBILITY:
Inclusion Criteria:

* Infants born in study communities who will reach 6 months of age during the six month period after initiation of the study

Exclusion Criteria:

* Infants likely to receive free or subsidized complementary foods (or infant formula)
* Families likely to relocate during the study period
* Infants with known congenital anomaly
* Infants of multiple birth
* Infants with neurological deficit apparent at the time of enrollment

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Stunting of Linear Growth | 18 months of age
  Stunting of linear growth will be defined as a height-for-age Z score less than 2 using WHO standards.

SECONDARY OUTCOMES:
Rate of Head Growth | 18 months of age
  Head circumference will be measured at enrollment (6 months of age) and conclusion of the study (18 months of age).
Incidence of wasting | 18 months of age
  Wasting will be defined as weight-for-age Z score less than 2 using the WHO growth standards.
Developmental Outcome | 18 months of age
  The Ages and Stages Questionnaire and the Bayley Scale of Infant Development II will be used to determine developmental outcome at 18 months of age.
Infectious Disease Morbidity | 6-18 months
  Infectious morbidities will be identified during weekly interviews of mothers by study personnel.
All Cause Mortality | 6-18 months
  Deaths will be reported to study personnel by family members or local health officials.
Compliance | 6-18 months
  Compliance with study protocol will be assessed by study personnel through interviewers with the mothers, direct observation, and recovery of unused cereal.
Iron Deficiency Anemia | 18 months
  We will measure serum markers of iron deficiency, including hemoglobin levels, ferritin and soluble transferrin receptor.

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Bose, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Kinshasa, Republic of the Congo

REFERENCES:
- [Derived] Bauserman M, Lokangaka A, Gado J, Close K, Wallace D, Kodondi KK, Tshefu A, Bose C. A cluster-randomized trial determining the efficacy of caterpillar cereal as a locally available and sustainable complementary food to prevent stunting and anaemia. Public Health Nutr. 2015 Jul;18(10):1785-92. doi: 10.1017/S1368980014003334. Epub 2015 Jan 29. PMID 25631295